CLINICAL TRIAL: NCT01961297
Title: Voice Tremor in Spasmodic Dysphonia: Central Mechanisms and Treatment Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kristina Simonyan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Kristina Simonyan, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 09-1156; R01DC012545 (NIH)
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Spasmodic Dysphonia; Voice Tremor
Keywords: dystonia; tremor; treatment; sodium oxybate; brain activity
MeSH Terms: conditions — Dysphonia; Dystonia; Tremor | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sodium oxybate (Experimental): Oral administration of a single dose of sodium oxybate (0.75-2.0 gm)
  Interventions: Drug: Sodium oxybate

INTERVENTIONS:
Drug: Sodium oxybate — Sodium oxybate
  Other Names: Xyrem

SUMMARY:
The proposed research aims to determine brain abnormalities in patients with spasmodic dysphonia (SD) and voice tremor (VT) as the basis for characterization of central mechanisms underlying symptom improvement following the use of sodium oxybate, a novel oral medication for the treatment of ethanol-responsive dystonia. The proposed research is relevant to public health because the elucidation of disorder-specific mechanistic aspects of brain organization in SD vs. SD/VT is ultimately expected to lead to establishment of enhanced criteria for clinical management of these disorders, including differential diagnosis and treatment. Thus, the proposed research is relevant to the part of NIH's mission that pertains to developing fundamental knowledge that will help to reduce the burdens of human disability.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD) is a chronic debilitating condition, characterized by selective loss of voluntary voice control during speech production due to uncontrolled spasms in the laryngeal muscles. SD becomes even more incapacitating when it is associated with action-induced voice tremor (VT) due to its poor response to gold standard treatment with botulinum toxin. There is, therefore, a critical need to identify new treatment opportunities for SD/VT patients who receive limited, if any, benefits from botulinum toxin injections. The design and use of novel therapeutic approaches for these patients will, however, be largely unattainable if the central mechanisms of SD and VT development remain unknown. Our long-term goal is to determine the pathophysiology of SD and related disorders, such as VT, for the development of new diagnostic and treatment options for these patients. The objective of this application is to identify brain abnormalities in SD and SD/VT patients as the basis for characterization of central mechanisms underlying symptom improvement following the use of sodium oxybate, a novel pharmacological agent for treatment of ethanol-responsive dystonia. Our central hypothesis is that, compared to SD patients, SD/VT patients will have additional brain abnormalities within the sensorimotor brain circuits controlling voice production, which are being modulated to a greater extent with sodium oxybate treatment. We further postulate that clinical efficacy of sodium oxybate treatment will correlate with its central modulatory effects. The rationale for the proposed research is that identification of distinct brain mechanisms underlying SD and SD/VT clinical manifestations would provide the necessary insights into the pathophysiology of these disorders, while understanding the neural correlates of sodium oxybate action would allow establishment of a scientific rationale for the use of a novel treatment in these disorders. Using a comprehensive approach of multi-modal neuroimaging and clinico-behavioral testing, our central hypothesis will be tested by pursuing two specific aims: (1) determine disorder-specific brain abnormalities in SD and SD/VT patients, and (2) characterize the central effects of sodium oxybate treatment in ethanol-responsive SD and SD/VT patients. This research is innovative because it focuses not only on identification of distinct pathophysiological factors contributing to SD and VT development, but also on discovery of mechanisms of central effects of a novel oral medication, sodium oxybate, which holds promise for treatment of refractory symptoms in SD and SD/VT. The proposed research is significant because it will advance our understanding of the pathophysiology of dystonia in general and SD in particular as well as will have direct impact on improvement of clinical management of SD and SD/VT patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented diagnosis of SD and/or VT with positive effects of alcohol on their symptoms;
* Age from 21 to 80 years;
* Native English speakers;
* Right-handedness (based on Edinburgh Handedness Inventory).

Exclusion Criteria:

* Subjects who are incapable of giving an informed consent;
* Pregnant and breastfeeding women until a time when they are no longer pregnant or breastfeeding will be excluded from the study. All patients of childbearing potential will be required to agree to use a reliable method of contraception prior and during the treatment with sodium oxybate and prior to receiving botulinum toxin. The method of contraception will be documented in the patient's research chart. All women of childbearing potential will undergo a urine pregnancy test, which must be negative for study participation;
* Subjects with past or present medical history of

  1. any neurological disorders, except for spasmodic dysphonia and voice tremor, will be excluded from the study in order to maintain the homogenous patient population, allow for the evaluation of drug effect on CNS without confounding by the presence of other neurological conditions, and identify SD and VT disorder-specific changes in brain function and structure. Patients who report other past or present neurological problems, such as stroke, movement disorders other than SD and VT, brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence will be excluded. As voice tremor is one of the forms of essential tremor, patients with moderate to severe essential tremor affecting other body parts will be excluded from the study. All patients who have dystonic movements in other than larynx body regions will also be excluded from the study;
  2. psychiatric problems, such as schizophrenia, major and/or bipolar depression, obsessive-compulsive disorder, will be excluded to maintain the homogenous patient population, allow for the evaluation of drug effect on CNS without confounding by the presence of psychiatric conditions and identify disorder-specific changes in brain function and structure;
  3. laryngeal problems, such as vocal fold paralysis, paresis, vocal fold nodules and polyps, carcinoma, chronic laryngitis;
  4. known past or present history of grade 2 or higher hepatic and renal dysfunction according to the NCI criteria.;
  5. known past or present history of moderate to severe congestive heart failure;
  6. known past or present history of cognitive impairment and active suicidal ideations;
* Patients who are not symptomatic due to treatment with botulinum toxin injections into the laryngeal muscles. The duration of positive effects of botulinum toxin vary from patient to patient but lasts on average for 3-4 months. All patients will be evaluated to ensure that they are fully symptomatic prior to the entering the study, except the substudy, which will examine the effects of combined botulinum toxin and sodium oxybate treatments on abnormal brain function in SD and VT patients;
* To avoid the possibility of confounding effects of drugs acting upon the central nervous system, all study participants will be questioned about any prescribed or over-the-counter medications as part of their initial intake screening. Those patients who receive medication(s) affecting the central nervous system (except sodium oxybate) will be excluded from the study.
* The participants will be asked whether they have undergone any head and neck surgeries, particularly any brain surgery and laryngeal surgeries, such as thyroplasty, laryngeal denervation, and selective laryngeal adductor denervation-reinnervation. Because both brain and laryngeal surgery may potentially lead to the brain structure and function re-organization, all subjects with history of brain and/or laryngeal surgery will be excluded from the study.
* The subjects who have tattoos, ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve, etc.) that cannot be removed for the purpose of MRI study participation.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Simonyan, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Simonyan K, Frucht SJ. Long-term Effect of Sodium Oxybate (Xyrem(R)) in Spasmodic Dysphonia with Vocal Tremor. Tremor Other Hyperkinet Mov (N Y). 2013 Dec 9;3:tre-03-206-4731-1. doi: 10.7916/D8CJ8C5S. eCollection 2013. PMID 24386608
- [Result] Rumbach AF, Blitzer A, Frucht SJ, Simonyan K. An open-label study of sodium oxybate in Spasmodic dysphonia. Laryngoscope. 2017 Jun;127(6):1402-1407. doi: 10.1002/lary.26381. Epub 2016 Nov 3. PMID 27808415
- [Derived] O'Flynn LC, Frucht SJ, Simonyan K. Sodium Oxybate in Alcohol-Responsive Essential Tremor of Voice: An Open-Label Phase II Study. Mov Disord. 2023 Oct;38(10):1936-1944. doi: 10.1002/mds.29529. Epub 2023 Jul 14. PMID 37448353
- [Derived] Simonyan K, Frucht SJ, Blitzer A, Sichani AH, Rumbach AF. A novel therapeutic agent, sodium oxybate, improves dystonic symptoms via reduced network-wide activity. Sci Rep. 2018 Oct 31;8(1):16111. doi: 10.1038/s41598-018-34553-x. PMID 30382161
- [Derived] Kirke DN, Frucht SJ, Simonyan K. Alcohol responsiveness in laryngeal dystonia: a survey study. J Neurol. 2015 Jun;262(6):1548-56. doi: 10.1007/s00415-015-7751-2. Epub 2015 May 1. PMID 25929664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 subjects were consented, some did not meet criteria, and 53 were enrolled into the study.
Groups:
- Spasmodic Dysphonia: Participants with Spasmodic Dysphonia (SD) given oral administration of a single dose of sodium oxybate (1.0-1.5 gm)
- Spasmodic Dysphonia/Voice Tremor: Participants with Spasmodic Dysphonia/Voice Tremor (SD/VT) given oral administration of a single dose of sodium oxybate (1.0-1.5 gm)
Period: Overall Study
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
Started | 30 | 23
Completed | 28 | 22
Not Completed | 2 | 1
Not completed — unconfirmed diagnosis of SD | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (11.3) | 58.0 (12.2) | 54.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 10 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 27 | 20 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Dystonia subtype [Count of Participants; unit: Participants] — ABSD = abductor spasmodic dysphonia; ADSD = adductor spasmodic dysphonia; VT = voice tremor
  Participants
    ADSD | 16 | 0 | 16
    ABSD | 12 | 0 | 12
    ADSD/VT | 0 | 15 | 15
    ABSD/VT | 0 | 7 | 7
Age of onset of dysphonia [Mean (Standard Deviation); unit: years] | 37.7 (11.0) | 44.1 (14.2) | 40.9 (12.6)
Duration of symptom of dysphonia [Mean (Standard Deviation); unit: years] | 13.4 (11.5) | 14.7 (12.7) | 14.1 (12.1)
Spasmodic dysphonia severity [Mean (Standard Deviation); unit: years] | 25.6 (16.3) | 30.3 (16.8) | 28.0 (16.6)
Voice Tremor severity [Mean (Standard Deviation); unit: units on a scale] — Only for participants that had voice tremor (VT). VT symptoms were evaluated using a visual analog scale of severity (0 for none, 100 for most severe/profound) Population: Only participants with voice tremor (VT)
  units on a scale
    number analyzed (Participants) | 0 | 22 | 22
    (all) |  | 49.3 (24.7) | 49.3 (24.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Positive Effects.
Description: Number of participants who had reported positive effects of at least one alcohol drink on their voice symptoms
Time Frame: Day 1
Population: Only alcohol-responsive participants were in this analysis which is 23 from the SD group and 22 from the SD/VT group.
Measure: Count of Participants; unit: Participants
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
Number analyzed (Participants) | 23 | 22
Participants | 17 | 20

2. Secondary Outcome: Number of Voice Breaks
Description: The number of SD-characteristic voice breaks in each sentence at pre-drug and post-drug assessment
Time Frame: baseline and Day 1
Population: Only alcohol-responsive participants were included in analysis
Measure: Mean (Standard Deviation); unit: voice breaks
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
Number analyzed (Participants) | 17 | 20
voice breaks
  Baseline - pre-treatment | 3.6 (1.6) | 4.1 (2.5)
  Day 1 - post treatment | 2.6 (1.8) | 2.8 (2.0)

3. Secondary Outcome: Voice Harshness Severity
Description: Visual analog scale of severity (0 for none, 100 for most severe/profound)
Time Frame: baseline and Day 1
Population: Only alcohol-responsive participants were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
Number analyzed (Participants) | 17 | 20
units on a scale
  Baseline - pre treatment | 48.0 (25.3) | 58.3 (23.1)
  Day 1 - post treatment | 42.8 (23.6) | 31.6 (17.8)

4. Secondary Outcome: Breathlessness Severity
Description: Visual analog scale of severity (0 for none, 100 for most severe/profound)
Time Frame: baseline and Day 1
Population: Only alcohol-responsive participants were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
Number analyzed (Participants) | 17 | 20
units on a scale
  Baseline - pre treatment | 24.0 (18.1) | 18.6 (25.2)
  Day 1 - post treatment | 20.0 (19.5) | 14.8 (19.2)

5. Secondary Outcome: Voice Tremor Severity
Description: Visual analog scale of severity (0 for none, 100 for most severe/profound)
Time Frame: baseline and Day 1
Population: Only alcohol-responsive participants with voice tremors were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
Number analyzed (Participants) | 0 | 20
units on a scale
  Baseline - pre treatment |  | 51.2 (23.6)
  Day 1 - post treatment |  | 31.4 (18.5)

ADVERSE EVENTS:
Time Frame: Up to 60 minutes after drug ingestion
Description: side effects questionnaire, Epworth Sleepiness Scale
Arm/Group | Spasmodic Dysphonia | Spasmodic Dysphonia/Voice Tremor
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 14/28 | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spasmodic Dysphonia (N=28) | Spasmodic Dysphonia/Voice Tremor (N=22)
Slight lightheadedness (Nervous system disorders) | 11 | 4
Drowsiness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
A limitation of this study was reliance on patients' self-reports of alcohol response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT01961297/Prot_SAP_000.pdf